CLINICAL TRIAL: NCT00486655
Title: Assisted Laparoscopic Cholecystectomy Surgery
Brief Title: NOTES-Assisted Laparoscopic Cholecystectomy Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of Focus for the company
Sponsor: USGI Medical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS0701
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Cholelithiasis; Cholecystitis
Keywords: Cholecystectomy; NOTES; Transgastric
MeSH Terms: conditions — Cholelithiasis; Cholecystitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: NOTES-Assisted Cholecystectomy

SUMMARY:
This study proposes to evaluate the ability to reduce the size and number of laparoscopic incisions required to perform gall bladder removal by using flexible endoscopic instruments introduced through the mouth, into the stomach and through the stomach wall.

DETAILED DESCRIPTION:
A typical laparoscopic gall bladder removal procedure requires placement of a rigid laparoscope through a 1.5-2.5 cm incision in the umbilicus and then 2-3 additional 0.5 cm incisions for additional instrumentation. While post-operative complication rates for this procedure are small, wound infection, particularly of the large incision, is one of the most common post-operative complications. There is also a risk of a post-operative hernia at these incision sites.

A less invasive surgical technique that reduces the size or number of laparoscopic incisions offers the potential clinical benefits of eliminating wound infections, hernias and decreasing post-operative pain following laparoscopic gall bladder removal.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo general anesthesia
* Age >= 18 yrs. of age and <= 85 yrs. of age
* Ability to give informed consent

Exclusion Criteria:

* Acute cholecystitis
* BMI >= 40
* Contraindicated for EGD
* Presence of common duct stones
* Presence of esophageal stricture
* Altered gastric anatomy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 2 weeks

SECONDARY OUTCOMES:
Incidence of complications | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lee Swanstrom, MD, Principal Investigator — Oregon Clinic
Locations (1):
- Oregon Clinic, Portland, Oregon, United States